CLINICAL TRIAL: NCT04421209
Title: Analgesic Effects of Perioperative Propranolol Administration for Spine Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding source
Sponsor: Duke University (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00103364
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Lumbar Disc Disease; Spinal Fusion; Degenerative Disc Disease
Keywords: lumbar fusion; propranolol; beta-blockers; post-surgical pain; opioid-sparing
MeSH Terms: conditions — Intervertebral disc disease; Intervertebral Disc Degeneration; Pain, Postoperative | interventions — Propranolol; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol treatment (Experimental): Subjects randomized to the propranolol treatment arm will be administered propranolol 40mg BID for three days prior to surgery, 40mg BID the day of surgery and on post-operative days 1 and 2. Subjects and researchers will be blinded and will not know if propranolol or placebo control is administered.
  Patients will be evaluated for opioid usend pain scores at 24 hrs, 48 hrs, 1 week, 4 weeks, and 12 weeks post-op.
  Blood will also be obtained pre-operatively, 8 hours and 24 hours post-operatively to measure the level of inflammatory markers. We will use these samples to evaluate if treatment with propranolol decreases the levels of inflammatory markers, and if this correlates to decreased opioid use and pain scores post-operatively.
  All other pre-, intra-, and post-operative interventions will be equivalent between the experimental and placebo groups, and this study's interventions will not affect surgical management.
  Interventions: Drug: Propranolol Hcl 40mg Tab
- Placebo (Placebo Comparator): Subjects randomized to the placebo treatment arm will be administered placebo tablets with the same schedule as propranolol in the experimental arm. Subjects and researchers will be blinded and will not know if propranolol or placebo control is administered.
  Patients will be evaluated for opioid use and pain scores at 24 hrs, 48 hrs, 1 week, 4 weeks, and 12 weeks post-op.
  Blood will also be obtained pre-operatively, 8 hours and 24 hours post-operatively to measure the level of inflammatory markers. We will use these samples to evaluate if treatment with propranolol decreases the levels of inflammatory markers compared to placebo, and if this correlates to decreased opioid use and pain scores post-operatively.
  All other pre-, intra-, and post-operative interventions will be equivalent between the experimental and placebo groups, and this study's interventions will not affect surgical management.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Propranolol Hcl 40mg Tab — 40mg PO BID for the three days prior to surgery, 40mg PO BID the day of surgery and on post-op days 1 and 2.
  Other Names: CAS No 525-66-6; DIN: 00496499; Inderal
  Arms: Propranolol treatment
Drug: Placebo oral tablet — Placebo tablets administered with the same schedule of Propranolol tablets
  Other Names: Tablet containing microcrystalline dextrose; Sugar pill, dextrose pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if treatment with low-dose oral propranolol in the days before and after surgery decrease postoperative pain and improve pain scores.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo controlled clinical trial.The main purpose of this study is to determine if postsurgical opioid use and pain scores are decreased with oral Propranolol treatment. The treatment period will last for six days and the observation period will last for three months. Effectiveness of treatment will be assessed by means of post-operative opioid consumption as primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age >18 undergoing elective spinal fusion surgery, with plans to remain inpatient for ≥ 48hrs and receive IV or oral opioids;
* Females of child bearing potential must test negative on a pregnancy test at Visit 1 and utilize acceptable means of birth control for the duration of the study;
* Patients must be judged by the study team to be likely to be reliable and to agree to keep all appointments for clinic visits, tests, and procedures required by the protocol;
* Patients must have the ability to fully participate in the informed consent process.

Exclusion Criteria:

* Disease-related: History of exercise- or exertion-induced asthma or current treatments for asthma; Unstable medical or neurological illness; Heart block greater than first degree (EKG); History of coronary artery disease, or history of congestive heart failure; Baseline heart rate or blood pressure that in the opinion of the investigator would constitute too great a risk when considered in the context of the patient's medical comorbidities and health history; Significant suicidal or homicidal ideation, or current DSM-IV diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, or cognitive disorder due to a general medical condition; History of diabetes
* Exposure-related: History of β-blocker use within six months of enrollment in the trial; Total baseline preoperative opioid consumption greater than 50 oral milligram morphine equivalents (MME) per day; Current use or use within the past two weeks of methadone, levorphanol, buprenorphine, butorphanol, pentazocine, tramadol, nalbuphine, naloxone, or naltrexone.
* Patient characteristics: Female patients who are pregnant or breast-feeding; Known allergy to study medication; Alcohol/substance abuse within past six months; Ongoing or anticipated disability compensation or litigation issues, in the best judgement of the investigator; Presence of any factors/conditions, medical or other, that in the judgment of the investigator may interfere with performance of study outcome measures, such as treatment-refractory history; Non-ambulatory or require the use of crutches or a walker; No access to a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative opioid use at 24 hours | 24 hours postoperatively
  Total opioid use from 0 to 24 hours post-op will be quantified. Opioid doses administered via all routes will be converted to standard oral morphine equivalents (OME).

SECONDARY OUTCOMES:
Acute postoperative opioid use at 48 hours | 48 hours postoperatively
  Total opioid use from 24 to 48 hours post-op will be quantified. Opioid doses administered via all routes will be converted to standard oral morphine equivalents (OME).
Sub-acute postoperative opioid use at 1 week | 1 week postoperatively
  Patient reported current opioid use for the prior 24 hours will be quantified at 1 week post-op. Opioid use will be converted to standard oral morphine equivalents (OME).
Sub-acute postoperative opioid use at 4 weeks | 4 weeks postoperatively
  Patient reported current opioid use for the prior 24 hours will be quantified at 4 weeks post-op. Opioid use will be converted to standard oral morphine equivalents (OME).
Sub-acute postoperative opioid use at 12 weeks | 12 weeks postoperatively
  Patient reported current opioid use for the prior 24 hours will be quantified at 12 weeks post-op. Opioid use will be converted to standard oral morphine equivalents (OME).
Acute postoperative pain scores at 24 hours | 24 hours post-op
  The CDC recommended 3-item Scale for Assessing Pain Intensity and Interference (PEG) will be used to assess postoperative pain over the past 24 hours. These data will be obtained at 24 post-op. The score is reported on a scale from 0 to 30. A higher score indicates more pain and therefore a worse outcome.
Acute postoperative pain scores at 48 hours | 48 hours post-op
  The CDC recommended 3-item Scale for Assessing Pain Intensity and Interference (PEG) will be used to assess postoperative pain over the past 24 hours. These data will be obtained at 48 hours post-op. The score is reported on a scale from 0 to 30. A higher score indicates more pain and therefore a worse outcome.
Sub-acute postoperative pain scores at 1 week | 1 week postoperatively
  The CDC recommended 3-item Scale for Assessing Pain Intensity and Interference (PEG) will be used to assess postoperative pain over the past 24 hours. These data will be obtained at 1 week post-op. The score is reported on a scale from 0 to 30. A higher score indicates more pain and therefore a worse outcome.
Sub-acute postoperative pain scores at 4 weeks | 4 weekspostoperatively
  The CDC recommended 3-item Scale for Assessing Pain Intensity and Interference (PEG) will be used to assess postoperative pain over the past 24 hours. These data will be obtained at 4 week post-op. The score is reported on a scale from 0 to 30. A higher score indicates more pain and therefore a worse outcome.
Sub-acute postoperative pain scores at 12 weeks | 12 weeks postoperatively
  The CDC recommended 3-item Scale for Assessing Pain Intensity and Interference (PEG) will be used to assess postoperative pain over the past 24 hours. These data will be obtained at 12 weeks post-op. The score is reported on a scale from 0 to 30. A higher score indicates more pain and therefore a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Buchheit, MD, Principal Investigator — Department of Anesthesiology, Duke University; Stephan Frangakis, MD/PhD, Study Director — Department of Anesthesiology, Duke University; William Maixner, DDS/PhD, Study Director — Department of Anesthesiology, Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afify EA, Andijani NM. Potentiation of Morphine-Induced Antinociception by Propranolol: The Involvement of Dopamine and GABA Systems. Front Pharmacol. 2017 Nov 10;8:794. doi: 10.3389/fphar.2017.00794. eCollection 2017. PMID 29209205
- [Background] Ciszek BP, O'Buckley SC, Nackley AG. Persistent Catechol-O-methyltransferase-dependent Pain Is Initiated by Peripheral beta-Adrenergic Receptors. Anesthesiology. 2016 May;124(5):1122-35. doi: 10.1097/ALN.0000000000001070. PMID 26950706
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Hartung JE, Ciszek BP, Nackley AG. beta2- and beta3-adrenergic receptors drive COMT-dependent pain by increasing production of nitric oxide and cytokines. Pain. 2014 Jul;155(7):1346-1355. doi: 10.1016/j.pain.2014.04.011. Epub 2014 Apr 13. PMID 24727346
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Krebs EE, Lorenz KA, Bair MJ, Damush TM, Wu J, Sutherland JM, Asch SM, Kroenke K. Development and initial validation of the PEG, a three-item scale assessing pain intensity and interference. J Gen Intern Med. 2009 Jun;24(6):733-8. doi: 10.1007/s11606-009-0981-1. Epub 2009 May 6. PMID 19418100
- [Background] Light KC, Bragdon EE, Grewen KM, Brownley KA, Girdler SS, Maixner W. Adrenergic dysregulation and pain with and without acute beta-blockade in women with fibromyalgia and temporomandibular disorder. J Pain. 2009 May;10(5):542-52. doi: 10.1016/j.jpain.2008.12.006. PMID 19411061
- [Background] Nackley AG, Tan KS, Fecho K, Flood P, Diatchenko L, Maixner W. Catechol-O-methyltransferase inhibition increases pain sensitivity through activation of both beta2- and beta3-adrenergic receptors. Pain. 2007 Apr;128(3):199-208. doi: 10.1016/j.pain.2006.09.022. Epub 2006 Nov 7. PMID 17084978
- [Background] Page MG, Kudrina I, Zomahoun HTV, Ziegler D, Beaulieu P, Charbonneau C, Cogan J, Daoust R, Martel MO, Neron A, Richebe P, Clarke H. Relative frequency and risk factors for long-term opioid therapy following surgery and trauma among adults: a systematic review protocol. Syst Rev. 2018 Jul 18;7(1):97. doi: 10.1186/s13643-018-0760-3. PMID 30021647
- [Background] Stanley TH, de Lange S, Boscoe MJ, de Bruijn N. The influence of chronic preoperative propranolol therapy on cardiovascular dynamics and narcotic requirements during operation in patients with coronary artery disease. Can Anaesth Soc J. 1982 Jul;29(4):319-24. doi: 10.1007/BF03007519. PMID 6213289
- [Background] Tchivileva IE, Lim PF, Smith SB, Slade GD, Diatchenko L, McLean SA, Maixner W. Effect of catechol-O-methyltransferase polymorphism on response to propranolol therapy in chronic musculoskeletal pain: a randomized, double-blind, placebo-controlled, crossover pilot study. Pharmacogenet Genomics. 2010 Apr;20(4):239-48. doi: 10.1097/FPC.0b013e328337f9ab. PMID 20216107
- [Background] Teimoori, B., Khoshfetrat, M., Beyrami, F., Sakhavar, N., Dehbashi, Z., Narouie, B., & Davarian, A. Propranolol decreases the post-operative pain and analgesic administration following abdominal hysterectomy. Life Sciences Journal 9: 1216-1220, 2012.
- [Background] Zanelatto FB, Dias EV, Teixeira JM, Sartori CR, Parada CA, Tambeli CH. Anti-inflammatory effects of propranolol in the temporomandibular joint of female rats and its contribution to antinociceptive action. Eur J Pain. 2018 Mar;22(3):572-582. doi: 10.1002/ejp.1143. Epub 2017 Dec 11. PMID 29226500